CLINICAL TRIAL: NCT00847067
Title: A Prospective, Single-blinded, Randomized, Trial Evaluating the Use of Paravertebral Block to Decrease Chronic Post Breast Surgery Pain.
Brief Title: Chronic Post Breast Surgery Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not renewed
Sponsor: Mayo Clinic (Other)
Responsible Party: Beth Ladlie, MD, Mayo Clinic Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 08-004783
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Block (Active Comparator)
  Interventions: Procedure: Paravertebral block
- Sham injection (Sham Comparator): Skin injections with Normal Saline
  Interventions: Procedure: Sham injections

INTERVENTIONS:
Procedure: Paravertebral block — 3ml 1% Ropivacaine at each level T1 - T5
  Arms: Block
Procedure: Sham injections — Sham injections with Normal Saline
  Arms: Sham injection

SUMMARY:
The purpose of this study is to learn if paravertebral block (PVB) will reduce chronic pain after surgery. Our hypothesis is that chronic pain from breast surgery as a consequence of central sensitization can be prevented by blocking sensory input to the CNS during surgery and the immediate post-operative period.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient who are ≥ 18 and ≤ 80 years of age.
2. Patient with diagnosis of breast cancer.
3. Patient scheduled for modified radical mastectomy or lumpectomy with axillary node dissection
4. Patient scheduled for one of the above listed surgeries with or without sentinel, partial, or complete axillary lymph node dissection
5. Patients scheduled for one of the aforementioned surgeries with or without immediate or delayed reconstruction.

Exclusion Criteria:

1. Pre-existing peripheral neuropathy
2. Pre-existing chronic pain
3. Bilateral procedure
4. Previous breast surgery, except biopsy
5. Inability to read, write or speak English.
6. Allergy to amide local anesthetics
7. Contraindications to paravertebral nerve block including, but not limited to severe scoliosis of the spine, skin lesion overlying the block area, abnormal coagulation studies (some of these may not be known until after informed consent is obtained)
8. Pregnancy
9. Emergency surgery
10. Previous recipients of peripheral nerve block.
11. Medical professional whose experience includes caring for patients who have had peripheral nerve blocks.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To obtain practical experience and information with which to develop a larger, more definitive study, particularly with regard to distributions of VAS responses at 3 months, patient compliance, and achievable accrual rate. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth Ladlie, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States